CLINICAL TRIAL: NCT01653028
Title: Phase II Study of MLN8237 in Advanced/Metastatic Sarcoma
Brief Title: Alisertib in Treating Patients With Advanced or Metastatic Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01991; NCI-2012-01991 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737403; A091102; CALGB-A091102; A091102 (Other: Alliance for Clinical Trials in Oncology); A091102 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Myxofibrosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Leiomyosarcoma; Recurrent Liposarcoma; Recurrent Malignant Peripheral Nerve Sheath Tumor; Recurrent Undifferentiated Pleomorphic Sarcoma; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7
MeSH Terms: conditions — Dermatofibrosarcoma; Sarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Histiocytoma, Malignant Fibrous | interventions — MLN 8237

ARMS (1):
- Treatment (alisertib) (Experimental): Patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well alisertib works in treating patients with sarcoma that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or has spread to other places in the body (metastatic). Alisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate (complete response [CR] + partial response [PR]) assessed for patients within each cohort: liposarcoma (cohort 1); leiomyosarcoma (non-uterine) (cohort 2); undifferentiated sarcoma (including pleomorphic undifferentiated sarcoma, formerly known as malignant fibrous histiocytoma, and myxofibrosarcoma) (cohort 3); malignant peripheral nerve sheath tumor (cohort 4); and other sarcomas (cohort 5).

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival (OS) for patients treated with MLN8237 (alisertib) in each cohort.

II. To assess the adverse events associated with patients treated with MLN8237 in each cohort.

TERTIARY OBJECTIVES:

I. To correlate potential clinical benefit with markers of aurora kinase inhibition in pre- and post-treatment tumor biopsies.

II. To correlate clinical outcome with change in fluorine F 18 fluorothymidine (FLT)-positron emission tomography (PET) uptake at baseline versus after one week of treatment (ie, week 2 of cycle 1).

OUTLINE:

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed sarcoma that is metastatic and/or locally advanced or locally recurrent and unresectable; confirmation of pathologic diagnosis will be performed at the registering site; patients will been rolled on one of five cohorts of the study:

  * Cohort 1: liposarcoma
  * Cohort 2: leiomyosarcoma (non-uterine)
  * Cohort 3: undifferentiated sarcoma (including malignant fibrous histiocytoma and myxofibrosarcoma)
  * Cohort 4: malignant peripheral nerve sheath tumor
  * Cohort 5: other sarcomas
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST) 1.1; note: defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 2 cm with conventional techniques or as >= 1 cm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Any number of prior therapies is permitted; note: the last dose of systemic therapy (including tyrosine kinase inhibitors) must have been given >= 4 weeks prior to initiation of study therapy; patients receiving BCNU or mitomycin C must have received their last dose of such therapy at least 6 weeks prior to initiation of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (alanine aminotransferase [AST]) < 3 x institutional upper limit of normal if no liver metastases or < 5 x institutional upper limit of normal if liver metastases present
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min/1.73m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MLN8237 administration
* Ability to understand and the willingness to sign a written informed consent document
* According to current guidelines, patients must be able to take oral medication and to maintain a fast as required for approximately one hour before and two hours after MLN8237 administration

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have had radiation therapy to more than 25% of the bone marrow; whole pelvic radiation is considered to be over 25%
* Patients who are receiving any other investigational agents
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN8237 including, but not limited to, established allergic reaction to benzodiazepines
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, New York Heart Association (NYHA) class II-IV heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women; note: women of child-bearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration; breastfeeding should be discontinued if the mother is treated with MLN8237
* Leiomyosarcoma of the uterus
* Patients known to be human immunodeficiency virus (HIV)-positive on antiretroviral therapy
* Prior allogeneic bone marrow or organ transplantation
* Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease, requirement for supplemental oxygen, or any conditions that could result in excessive toxicity associated with the benzodiazepine-like effects of MLN8237
* Requirement for constant administration of proton pump inhibitor, histamine-2 (H2) antagonist, or pancreatic enzymes; note: intermittent uses of antacids or H2 antagonists are allowed
* Inability to swallow oral medication or to maintain a required fast for approximately one hour before and two hours after MLN8237 administration or any condition that would modify small bowel absorption of oral medications, including malabsorption or resection of pancreas or upper bowel
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, oxcarbazepine, primidone or phenobarbital, or rifampin, rifabutin, rifapentine, or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2015-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dickson, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (235):
- United States (235):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Kootenai Cancer Center, Post Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Dickson MA, Mahoney MR, Tap WD, D'Angelo SP, Keohan ML, Van Tine BA, Agulnik M, Horvath LE, Nair JS, Schwartz GK. Phase II study of MLN8237 (Alisertib) in advanced/metastatic sarcoma. Ann Oncol. 2016 Oct;27(10):1855-60. doi: 10.1093/annonc/mdw281. Epub 2016 Aug 8. PMID 27502708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2012 to April 2014, a total of 72 patients were accrued to this study (Cohort 1 - 12, Cohort 2 - 10, Cohort 3 - 11, Cohort 4 - 10 Cohort 5 - 29) at a rate of 4.5 patients per month.
Groups:
- Cohort 1: Liposarcoma patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cohort 2: Leiomyosarcoma patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cohort 3: Undifferentiated Sarcoma patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cohort4: Malignant Peripheral Nerve Sheath Tumor patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Cohort 5: Other Sarcoma patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort4 | Cohort 5
Started | 12 | 10 | 11 | 10 | 29
Completed | 12 | 10 | 11 | 10 | 29
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort4 | Cohort 5 | Total
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 29 | 72
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 72] | 56.5 [39 to 84] | 66 [49 to 76] | 52.5 [29 to 71] | 49 [20 to 83] | 54.5 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 5 | 4 | 14 | 33
  Male | 5 | 7 | 6 | 6 | 15 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 2 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2 | 2 | 6
  White | 10 | 10 | 9 | 7 | 25 | 61
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 11 | 10 | 29 | 72

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint for This Trial Was the Percent of Confirmed Tumor Responses. Confirmed Tumor Response to Treatment Was Defined as a Complete or Partial Response(Per RECIST 1.1) on Two Consecutive Evaluations at Least 6 Weeks Apart.
Description: The primary endpoint was estimated by the number of confirmed responses divided by the total number of evaluable patients per cohort. The study used a two stage Simon design to assess the primary endpoint. A confirmed tumor response rate of 5% was considered not promising; an observed confirmed response rate of 25% was considered promising. One confirmed response within the initial 9 patients enrolled within each cohort, expanded enrollment to 24 patients in that cohort. 3 out of 24 patients with confirmed tumor responses was considered evidence that this treatment could be recommended for further testing. This study design yielded 90% power to detect a true confirmed response rate of at least 25% at .10 level of significance if the true rate is at most 5%. There was a 63% chance of stopping early if the true confirmed response rate was 5%.
Time Frame: Up to 18 months
Measure: Number; unit: percentage of patients with response
Groups:
- Cohort 4: Malignant Peripheral Nerve Sheath Tumor patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 29
percentage of patients with response | 0 | 0 | 0 | 0 | 7

2. Secondary Outcome: Overall Survival (OS)
Description: The distribution will be estimated by the methods of Kaplan and Meier. The estimates of survival at specific time points will be calculated (eg, median, 6 month survival).
Time Frame: The time between registration and death, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 29
Weeks | NA [23.3 to NA] — Not Reached | 71.7 [16 to NA] — Not Reached | 67.8 [19 to NA] — Not Reached | 69 [16 to NA] — Not Reached | 28.6 [16.6 to 51.3]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The distribution will be estimated by the methods of Kaplan and Meier. The estimates of PFS at specific time points will be calculated (eg, median, 1 year PFS).
Time Frame: The time between registration to disease progression or death, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 29
Weeks | 13 [6.29 to 37.1] | 11.7 [1.71 to 21.9] | 11.7 [5 to 20.6] | 13.2 [3.57 to 45] | 6.57 [5.86 to 18.1]

4. Secondary Outcome: Adverse Events
Description: Adverse Events: Incidence of adverse events, assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Adverse events were collected every cycle during treatment and up to one month after treatment. Adverse events were summarized using summary statistics and frequency tables for each separate cohort. Per protocol, analysis was descriptive in nature. In this section, the number of patients that reported a grade 4 or higher event are summarized. A complete listing of Adverse Events is provided in the Adverse Events section below.
Time Frame: During treatment and up to 5 years
Population: All patients that began study treatment were assessed for this endpoint.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 10 | 11 | 10 | 29
participants
  Grade 4 Event | 6 | 1 | 5 | 0 | 4
  Grade 5 Event | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort4 | Cohort 5
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/10 | 1/11 | 4/10 | 13/29
Other Adverse Events (participants affected / at risk) | 12/12 | 8/10 | 11/11 | 9/10 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=10) | Cohort 3 (N=11) | Cohort4 (N=10) | Cohort 5 (N=29)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=10) | Cohort 3 (N=11) | Cohort4 (N=10) | Cohort 5 (N=29)
Anemia (Blood and lymphatic system disorders) | 10 (32) | 4 (15) | 7 (44) | 6 (15) | 15 (37)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dry eye (Eye disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (2) | 0 (0) | 1 (2)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (4) | 1 (2) | 3 (3) | 3 (12)
Diarrhea (Gastrointestinal disorders) | 4 (9) | 2 (5) | 4 (15) | 6 (16) | 11 (28)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (6) | 4 (4) | 4 (5) | 5 (8) | 11 (28)
Nausea (Gastrointestinal disorders) | 6 (27) | 1 (2) | 4 (11) | 5 (7) | 7 (24)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (9) | 0 (0) | 2 (2) | 2 (2) | 3 (7)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 10 (42) | 6 (16) | 4 (12) | 6 (12) | 13 (39)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 1 (4) | 2 (2) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (11) | 4 (4) | 2 (22) | 4 (5) | 7 (23)
Neutrophil count decreased (Investigations) | 6 (26) | 5 (9) | 8 (20) | 5 (7) | 17 (41)
Platelet count decreased (Investigations) | 5 (29) | 5 (15) | 6 (19) | 3 (5) | 14 (66)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 7 (35) | 4 (6) | 6 (38) | 6 (9) | 12 (45)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 2 (8) | 2 (2) | 4 (21)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 3 (12) | 3 (7) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (11) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (7)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2) | 3 (6) | 4 (6) | 7 (15)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (4) | 3 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (6) | 1 (5) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (37) | 4 (19) | 8 (44) | 8 (24) | 17 (79)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (10) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 4 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (22) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 1 (4) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less